CLINICAL TRIAL: NCT05290350
Title: Obstructive Sleep Apnea in Patients With Long COVID-19 Fatigue: a Multicentre Prospective Cohort Study
Brief Title: Long COVID-19 Fatigue and Obstructive Sleep Apnea
Acronym: PostCoV2OSA
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Centro Hospitalar Universitario do Algarve (Other)
Collaborators: Sociedade Portuguesa de Pneumologia (Other); Universidade do Algarve (Other); Universidade do Porto (Other); Center for Health Technology and Services Research (Other); Linde Health Care (Other)
Responsible Party: Principal Investigator, Ligia Pires, Principal Investigator, Centro Hospitalar Universitario do Algarve
Other Study IDs: 132/21
Record Dates: First submitted 2022-03-19; First posted 2022-03-22 (Actual); Last update posted 2022-04-06 (Actual); Status verified 2022-03

CONDITIONS: Long COVID; Fatigue; Obstructive Sleep Apnea of Adult
Keywords: Post-COVID-19 fatigue Sleep Apnea SARS-CoV-2 Vaccines
MeSH Terms: conditions — Post-Acute COVID-19 Syndrome; Fatigue

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- OSA Cohort: Patients With post COVID-19 condition and OSA
  Interventions: Other: OSA
- Control Cohort: Patients With post COVID-19 condition without OSA

INTERVENTIONS:
Other: OSA — EXPOSURE TO OBSTRUCTIVE SLEEP APNEA
  Groups: OSA Cohort

SUMMARY:
Identify the relationship of obstructive sleep apnea (OSA) prevalence with post-COVID-19 fatigue that remains at least six months after acute disease

DETAILED DESCRIPTION:
The presence of fatigue symptoms up to 6-7 months after acute COVID-19 disease, similar to myalgic encephalomyelitis/chronic fatigue syndrome, also observed after other viral infections, have been reported as the most frequent post-COVID-19 symptom (Townsend et al., 2020).

There is a physiological plausibility for OSA being a causal factor to COVID-19 morbidity and fatigue symptoms by nocturnal hypoxemia, exacerbating or causing endothelial dysfunction, inflammation, oxidative stress, microaspiration and cardiac dysfunction. OSA activates the renin-angiotensin-aldosterone system (RAAS) and angiotensin-converting enzyme-2 (ACE2), which is the SARS-CoV-2 entry receptor in the cells (Miller et al., 2021).

In this study we will identify the prevalence of OSA and it's relation with post-COVID-19 fatigue that remains for at least six month after the acute disease, in patients that attend the post-COVID-19 Out Patients Hospital Clinics. It will be studied also the relation between fatigue and vaccination status, nocturnal hypoxemia, day time sleepness and the acute COVID-19 severity.

Data collection will be performed by a questionnaire administered by qualified clinical study staff (i.e., by physicians who conduct the post-COVID-19 medical consultation).

Demographic, clinical data and clinical research forms will be collected between 6-7th month after the diagnosis of COVID-19 (t1) and 9 months later (t2).

Fatigue will be assessed using the Chalder fatigue scale - CFQ-11 (Chalter et al., 1993).

The evaluation of OSA related daytime sleepiness will be measured using the Epworth Sleepiness Scale - ESS (Johns, 1991). The OSA diagnosis will be performed using portable monitoring device type III (in-home polygraphy), between 6-7th month after the diagnosis of COVID-19 (t1).

ELIGIBILITY:
Inclusion Criteria:

(1) ≥18 years; (2) previous COVID-19 at least six months before the initial study protocol evaluation; (3) persistent symptoms after cure criteria defined by WHO; (4) patients who attend the post-COVID-19 follow-up consultation of the study centers. (5) SARS-CoV-2 infection confirmed by a positive real-time reverse-transcription polymerase chain reaction on a nasopharyngeal swab (6) patients who agree to sign the Written informed consent (following the ethics committee protocol).

Exclusion Criteria:

(1) patients who had a concomitant neurological disorder that could increase OSA risk (such as stroke, Parkinson disease, or amyotrophic lateral sclerosis); (2) patients who were on invasive mechanical ventilation. (3) patients with persistent fatigue symptoms,6 months before SARS-CoV-2 infection (4) patients without SARS-CoV-2 positive real-time reverse-transcription polymerase chain reaction on a nasopharyngeal swab

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study will be conducted in twelve Portuguese Hospitals, Universitary and District, in which a follow-up post-COVID-19 medical consultation has been implemented All patients that attend the follow-up post COVID-19 consultation will be invited to participate in the study.
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2022-03-10 (Actual); Primary Completion 2022-11-30 (Estimated); Study Completion 2023-01-30 (Estimated)

PRIMARY OUTCOMES:
post-COVID-19 long term fatigue and OSA | 6 - 7 months
  Evaluate if untreated OSA is associated with post COVID-19 long term fatigue.

SECONDARY OUTCOMES:
post-COVID-19 long term fatigue and daytime sleepiness | 6 - 9 months
  Evaluate if daytime sleepiness is associated with post COVID-19 long term fatigue.
post-COVID-19 long term fatigue and nocturnal hypoxemia | 6 - 7 months
  Evaluate if nocturnal hypoxemia is associated with post COVID-19 long term fatigue
post-COVID-19 long term fatigue and severity of acute COVID-19 | 6 - 9 months
  Evaluate if severity of acute COVID-19 is associated with post COVID-19 long term fatigue
post-COVID-19 long term fatigue and vaccination status | 6 - 9 months
  Study the relation between vaccination status and post-COVID-19 long term fatigue
Long COVID-19 and OSA impact in quality of life | 6 - 7 months
  Study the impact of Long COVID-19 with untreated OSA in quality of life

CONTACTS AND LOCATIONS:
Overall Officials: Ligia Pires, Study Chair — Centro Hospitalar Universitario do Algarve
Locations (12):
- Portugal (12):
  - Hospital Particular de Alvor, Alvor
  - Hospital de Faro (Chua), Faro
  - Hospital da Luz Guimaraes (HLG), Guimarães
  - Hospital de Santo Andre (Chl), Leiria
  - Hospital Da Luz Lisboa, Lisbon
  - Hospital de Santa Maria (CHULN), Lisbon
  - Hospital Beatriz Angelo (Hba), Loures
  - Hospital de Portimao (Chua), Portimão
  - Hospital Sao Joao (Chusj), Porto
  - Hospital de Sao Sebastiao (Chedv), Santa Maria da Feira
  - Centro Hospitalar de Setubal (Chs), Setúbal
  - Centro Hospitalar De Trás-Os-Montes E Alto Douro (CHTMAD), Vila Real

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Chalder T, Berelowitz G, Pawlikowska T, Watts L, Wessely S, Wright D, Wallace EP. Development of a fatigue scale. J Psychosom Res. 1993;37(2):147-53. doi: 10.1016/0022-3999(93)90081-p. PMID 8463991
- [Background] Johns MW. A new method for measuring daytime sleepiness: the Epworth sleepiness scale. Sleep. 1991 Dec;14(6):540-5. doi: 10.1093/sleep/14.6.540. PMID 1798888
- [Background] Miller MA, Cappuccio FP. A systematic review of COVID-19 and obstructive sleep apnoea. Sleep Med Rev. 2021 Feb;55:101382. doi: 10.1016/j.smrv.2020.101382. Epub 2020 Sep 8. PMID 32980614
- [Background] Townsend L, Dyer AH, Jones K, Dunne J, Mooney A, Gaffney F, O'Connor L, Leavy D, O'Brien K, Dowds J, Sugrue JA, Hopkins D, Martin-Loeches I, Ni Cheallaigh C, Nadarajan P, McLaughlin AM, Bourke NM, Bergin C, O'Farrelly C, Bannan C, Conlon N. Persistent fatigue following SARS-CoV-2 infection is common and independent of severity of initial infection. PLoS One. 2020 Nov 9;15(11):e0240784. doi: 10.1371/journal.pone.0240784. eCollection 2020. PMID 33166287